CLINICAL TRIAL: NCT02035423
Title: Community Interventional Trial (CITFOMIST) to Study the Efficacy and Compliance of Different Degrees of Vitamin D Fortified Milk
Brief Title: Community Interventional Trial (CITFOMIST)
Acronym: CITFOMIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EMRI-1390; CITFOMIST (Other: EMRI)
Record Dates: First submitted 2013-12-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency; Compliance; Milk
MeSH Terms: conditions — Vitamin D Deficiency; Patient Compliance | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Male Guidance School (Active Comparator): Non-Fortified Milk 120IU Milk 200IU Milk
  Interventions: Dietary Supplement: 120 IU milk; Dietary Supplement: 200 IU Milk; Dietary Supplement: Non-Fortified Milk
- Female Guidance (Active Comparator): Non-fortified Milk 120IU Milk 200IU Milk
  Interventions: Dietary Supplement: 120 IU milk; Dietary Supplement: 200 IU Milk; Dietary Supplement: Non-Fortified Milk
- Male Highschool (Active Comparator): Non-Fortified Milk 120IU Milk 200IU Milk
  Interventions: Dietary Supplement: 120 IU milk; Dietary Supplement: 200 IU Milk; Dietary Supplement: Non-Fortified Milk
- Female Highschool (Active Comparator): Non-Fortified Milk 120IU Milk 200IU Milk
  Interventions: Dietary Supplement: 120 IU milk; Dietary Supplement: 200 IU Milk; Dietary Supplement: Non-Fortified Milk

INTERVENTIONS:
Dietary Supplement: 120 IU milk — Daily consumption of milk fortified with 120 IU vitamin D
Dietary Supplement: 200 IU Milk — Daily Consumption of milk fortified with 200 IU vitamin D
Dietary Supplement: Non-Fortified Milk — Daily consumption of non-fortified milk

SUMMARY:
The cluster randomized trial (CITFOMIST) was conducted on 15-19-year old guidance and high school students of both genders from different districts of Tehran, the Iranian capital, in winter 2011. The 36 schools enrolled in this study were randomly assigned to receive one of the three groups of milk -- whole milk, milk that contained 600 IU Vit D/1000cc, milk that contained 1000 IU Vit D /1000cc -- for a 30-day period. In order to study the effect of vitamin D-fortified milk on the circulating concentrations of 25(OH)D, a serum vitamin D levels were checked in a subgroup before and after the intervention.

DETAILED DESCRIPTION:
The cluster randomized trial (CITFOMIST) was conducted on 15-19-year old guidance and high school students of both genders from different districts of Tehran, the Iranian capital, in winter 2011.

The 36 schools enrolled in this study were randomly assigned to receive one of the three groups of milk -- whole milk, milk that contained 600 international unit (IU) Vit D/1000cc (120IU), milk that contained 1000 IU Vit D /1000cc (200IU)-- for a 30-day period. In order to study the effect of vitamin D-fortified milk on the circulating concentrations of 25(OH)D, a serum vitamin D levels were checked in a subgroup before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 15-19-year old guidance and high school students of both genders from different districts of Tehran, the Iranian capital

Exclusion Criteria:

* Those taking vitamin D supplements
* Those with underlying disease affecting bone health
* Those taking medication affecting bone metabolism
* Those taking fortified products on a regular basis
* Those following special diets

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6000 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Compliance with milk consumption | 1 month

SECONDARY OUTCOMES:
Serum 25(OH)D levels | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Khashayar, Principal Investigator — Endocrinology and Metabolism Research Institute; Abbasali Keshtkar, Study Director — Endocrinology and Metabolism Research Institute; Bagher Larijani, Study Chair — Endocrinology and Metabolism Research Institute
Locations (1):
- EMRI, Tehran, Iran